CLINICAL TRIAL: NCT01418482
Title: An Open Non-controlled Post-marketing Investigation Evaluating the Experience of Using a Self- Adherent Antimicrobial Soft Silicone, Silver Containing, Foam Dressing, Mepilex Border Ag, in Second Degree Burns
Brief Title: Evaluation of Antimicrobial Soft Silicone, Silver Containing, Foam Dressing, Mepilex Border Ag, in Second Degree Burns
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Molnlycke Health Care AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MxB Ag 02
Record Dates: First submitted 2011-01-27; First posted 2011-08-17 (Estimated); Results first posted 2017-05-03 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2011-08

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mepilex Border Ag (Experimental): Mepilex Border Ag, a silver dressing will be used
  Interventions: Device: Mepilex Border Ag

INTERVENTIONS:
Device: Mepilex Border Ag — a silver dressing

SUMMARY:
The investigation is designed as an open, non-controlled, post-marketing investigation. Subjects with at least one second degree burn less than 9.5x15 cm in size at 1-3 sites will be included. The subject is allowed to have more than one burn on the body but only one should be included in the investigation. Each subject will be followed/assessed according to normal hospital routine 1-3 times per week for a maximum of 3 weeks or until desired treatment effect is obtained if that occurs earlier. All dressing changes will be done according to clinical routine and will follow the IFU (instruction for use). All dressing changes will be registered in a dressing log. Additional compression bandaging, gauze wrap, or such are allowed and should be reported as well

DETAILED DESCRIPTION:
At baseline, subject characteristics will be registered together with subject status of health and status of the burn, and current treatment of the burn.

At each visit the following variables will be collected where applicable:

* Investigator's/Nurse evaluation of

  * Overall experience of the dressing
  * Ability of dressing to stay in place (not at baseline)
  * Conformability of the dressing
  * Handling at application
  * Ease of removal of the dressing (not at baseline)
* Subject evaluation of

  * Overall experience of the dressing
  * Comfort of the dressing
  * Conformability of the dressing
* Pain before, during and after removal of dressing according to VAS
* Status of skin
* Burn status: width x length, exudate details and signs of inflammation/infection

In addition the following variables should be evaluated at each visit:

* Concomitant medication/treatment
* Adverse Event/Adverse Device Effect (AE/ADE)
* Serious Adverse Event/Serious Adverse Device Effect (sAE/sADE)

Photos will be taken before Mepilex Border Ag is removed, after removal, before cleansing, and after cleansing. All photos must include a sticker marker with subject code, visit number and date, and an indication of whether pre-/post removal, pre-/post cleansing. The stick marker also contains a ruler. Detailed instructions on how to take the photos is given in Appendix 14.2

At each visit the subject will give the assessment concerning the comfort and stay-on-ability of the dressing. The investigator will also give an assessment at each visit concerning handling, conformability and ability of dressing to stay in place.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with a small partial thickness burn (< 9.5x15 cm) where an antimicrobial action is indicated as judged by the investigator*
2. Male or female, 18 years and above, both in- and out-patient subjects
3. Signed Informed Consent Form

Exclusion Criteria:

1. Wound size equal to or above 9.5x15cm for the selected burn for the investigation
2. Pregnant and/or breastfeeding women
3. Subject not expected to follow the investigation procedures or applicable for investigation according to the judgment of the investigator
4. Subjects with known sensitivity to silver or any other contents of the dressing
5. Subjects previously included in this investigation
6. Subjects included in other ongoing clinical investigation at present or during the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-01; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik Huss, MD, Principal Investigator — Akademiska Hospital
Locations (2):
- Sweden (2):
  - Briva/Hpk, Linköping
  - Plastikkirurgiska kliniken, UAS BRIVA, Uppsala

RESULTS

PARTICIPANT FLOW:
Groups:
- Mepilex Border Ag: Mepilex Border Ag, a silver dressing
Period: Overall Study
Arm/Group | Mepilex Border Ag
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: small partial thickness burns
Groups:
- Mepilex Border Ag: Mepilex Border Ag, ( a silver dressing)
Arm/Group | Mepilex Border Ag
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Region of Enrollment [Number; unit: participants]
  Sweden | 15

OUTCOME MEASURES:

1. Primary Outcome: Evaluate the Experience of Using Mepilex Border Ag ( a Silver Dressing) in Normal Clinical Practice
Description: burns healed
Time Frame: 3 weeks
Population: small thickness partial burns
Measure: Number; unit: burns healed
Groups:
- Mepilex Border Ag: Mepilex Border Ag
Arm/Group | Mepilex Border Ag
Number analyzed (Participants) | 15
burns healed | 9

2. Secondary Outcome: Evaluate the Comfort
Description: Comfort level and overall experience were each assessed using a scale that ranged from very poor to very good.
Time Frame: 3 weeks
Measure: Number; unit: participants
Arm/Group | Mepilex Border Ag
Number analyzed (Participants) | 15
participants
  Conformability Good -very Good | 15
  Overall experience good-very good | 14

3. Secondary Outcome: Pain
Description: To evaluate pain during dressing removal at visit 4,(after one week) with John Hopkins pain scale. Measured 0=no pain, 100= worst pain, scale from 0-100 mm
Time Frame: 3 weeks
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Mepilex Border Ag
Number analyzed (Participants) | 15
units on a scale | 0 [0 to 40]

ADVERSE EVENTS:
Arm/Group | Mepilex Border Ag
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 2/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mepilex Border Ag (N=15)
Swelling of left hand (General disorders) | 1 (1) — Swelling of left hand
Infection left arm, no study burn (Infections and infestations) | 1 (1) — Infection left arm, no study burn

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less